CLINICAL TRIAL: NCT00948844
Title: Automatic Detection of Falls and Near Falls
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Jeffrey Hausdorff, PhD, Director of gait lab, Tel-Aviv Sourasky Medical Center
Other Study IDs: TASMC - 09 - NG - 521 - CTIL
Record Dates: First submitted 2009-05-27; First posted 2009-07-29 (Estimated); Last update posted 2009-07-29 (Estimated); Status verified 2009-07

CONDITIONS: Falls; Missteps
Keywords: falls; Missteps

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Hybrid (3-d accelerometers, and gyroscopes) — A 3 D accelerometer worn on the lower back or leg
  Other Names: McRoberts

SUMMARY:
The aim of this study is to develop an algorithm to automatically detect falls and near falls, in the elderly and in Parkinson's Disease patients. Subjects will arrive at the investigators' gait laboratory for assessment. A sub-group of the subjects, will receive a monitoring device, to be worn at home for three days.

DETAILED DESCRIPTION:
The aim of this study is to develop a detailed algorithm which will automatically detect falls and near falls, in the elderly as a general population prone to falls. The algorithm will be used as well in patients with Parkinson's Disease representing neurodegenerative diseases. All participants will arrive at the investigators' gait laboratory for an inhanced assessment, including neurological examination, various questionnaires. A sub-group of the subjects, will receive a monitoring device, to be worn at home for three days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Older Adults
* Parkinson's Disease Patients
* Idiopathic Fallers

Exclusion Criteria:

* Walking Aid
* Other Neurological Diseases than PD
* Significant Disturbance in Vision/Hearing
* History of CVA
* Significant Orthopedic Problem
* Dementia

Ages: 50 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Healthy Older Adults
  * Parkinson's Disease Patients
  * Idiopathic Fallers
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2009-08; Primary Completion 2010-08 (Estimated); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
3 D acceleration | during assessment

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey M Hausdorff, PhD, Study Director — Tel-Aviv Sourasky Medical Center
Locations (1):
- Labrotory for Gait and Neurodynamics, Movement Disorders Unit, TASMC, Tel Aviv, IL, Israel